CLINICAL TRIAL: NCT05303025
Title: Qualitative Research Among Physicians and Junior Doctors Into the Preconditions for Implementing a Clinical Decision Support System (CDSS) Based on Artificial Intelligence (AI) in the ICU
Brief Title: Qualitative Research Among Physicians and Junior Doctors Into the Preconditions for Implementing a CDSS Based on AI in the ICU
Acronym: KATRINA
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Sponsor
Other Study IDs: BC-9892
Record Dates: First submitted 2022-02-22; First posted 2022-03-31 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2022-10

CONDITIONS: Artificial Intelligence; Qualitative Research; Decision Support Systems, Clinical
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Survey to acquire baseline demographic information as well as information regarding professional experience, working environment and attitudes towards artificial intelligence.
Other: Semi-structured group discussion — Semi-structured group discussion.

SUMMARY:
The goal of this study is to explore the different attitudes and preconditions of potential end-users (doctors & physicians in training) required to achieve successful clinical implementation of models based on artificial intelligence (i.e. both machine learning and knowledge-driven techniques) as clinical decision support software.

ELIGIBILITY:
Inclusion Criteria:

* Medical specialist or specialist in training working in intensive care at the time of the study.

Exclusion Criteria:

* Age < 18 yo

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical specialists or specialists in training working in intensive care at the time of the study.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Baseline attitudes towards artificial intelligence and big data in medicine | baseline
  Baseline attitudes towards artificial intelligence and big data in medicine will be collected through an online survey where participants will score their agreement with certain statements on a 6-point likert scale (Possible choices: Strongly agree - Agree - Neutral - Disagree - Totally Disagree - Not applicable).
Identify subdomains of the antimicrobial stewardship cycle with potential for AI/Big data application | through study completion, an average of 1 year
  Identify subdomains of the antimicrobial stewardship cycle for which participants think AI/Big data might be of use through a group discussion/interview. Reporting: frequencies.
Identify perceived potential benefits and harms when applying AI in the antimicrobial stewardship cycle. | through study completion, an average of 1 year
  Identify perceived potential benefits and harms when applying AI in the antimicrobial stewardship cycle through a group discussion. Reporting: frequencies.
Identify prerequisites that need to be fulfilled when AI/Big data based clinical decision support systems are used bedside from the viewpoint of the participants. | through study completion, an average of 1 year
  Identify prerequisites that need to be fulfilled when AI/Big data based clinical decision support systems are used bedside and identify the most important ones for different aspects of the antimicrobial stewardship cycle from the viewpoint of the participants through a group discussion. Reporting: frequencies.

SECONDARY OUTCOMES:
Subgroup analysis: age | through study completion, an average of 1 year
  Explore if there are variations in the above mentioned outcomes when taking into account the age (years) of the participants.
Subgroup analysis: gender | through study completion, an average of 1 year
  Explore if there are variations in the above mentioned outcomes when taking into account the gender of the participants.
Subgroup analysis: working environment (type of hospital, type of ICU) | through study completion, an average of 1 year
  Explore if there are variations in the above mentioned outcomes when taking into account the working environment (University hospital vs non University hospital, small size hospital vs large size hospital, type of ICU (medical, surgery, mixed ICU, intermediate care)) - data which is collected in the baseline questionnaire) of the participants.
Subgroup analysis: working experience (basic training and clinical experience). | through study completion, an average of 1 year
  Explore if there are variations in the above mentioned outcomes when taking into account the working experience (type of basic training (anesthesiology, internal medicine, surgery, other), clinical experience (years) - data which is collected in the baseline questionnaire) of the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Jan De Waele, MD, PhD, Principal Investigator — University Ghent
Locations (3):
- Belgium (3):
  - OLV Aalst, Aalst
  - ZNA Ziekenhuizen, Antwerp
  - Ghent University Hospital, Ghent

IPD SHARING:
Plan to Share IPD: Undecided
If possible and feasible, anonymised survey data as well as transcript data from the group discussions will be made available on request.